CLINICAL TRIAL: NCT01637948
Title: Controlled Clinical Trial of Traditional Chinese Medicine Mouthrinse In Improving Oral Health in Orthodontic Patients
Brief Title: Controlled Clinical Trial of Traditional Chinese Medicine Mouthrinse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Wing Kit, Ricky, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-1145
Record Dates: First submitted 2012-01-03; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Gingivitis
Keywords: Chinese medicine; gingivitis; cytokine; microbial
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Listerine (Active Comparator): essential oil mouthrinse
  Interventions: Drug: Listerine mouthrinse
- Negative control (No Intervention): without intervention
- Chinese medicine mouthrinse (Experimental): 5% Fructus Mume extract and 2% sodium bicarbonate
  Interventions: Drug: Chinese Medicine mouthrinse

INTERVENTIONS:
Drug: Listerine mouthrinse — For six months
  Other Names: essential oils mouthrinse
  Arms: Listerine
Drug: Chinese Medicine mouthrinse — six months
  Other Names: 5% Fructus mume and 2% soudium bicarbonate
  Arms: Chinese medicine mouthrinse

SUMMARY:
Traditional Chinese medicine (TCM) has been seen as the predominant way of treating disease in China over three thousand years. Certain TCM have scientifically proved to have anti-bacterial property. Patients having orthodontic treatment have higher risks of caries and gum diseases. The purpose of this study was to determine whether the use of TCM Mouthrinses in addition to toothbrushing and flossing has an added benefit for orthodontic patients in maintaining proper oral health.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of a Traditional Chinese medicine (TCM) mouthrinse on gingival health and microbial profiles in orthodontic patients. This six-month randomized, single-blinded, parallel controlled clinical trial consists of 90 patients with fixed appliance treatment. The subjects were allocated to (1) negative-control group: oral hygiene instruction (OHI) alone; (2) positive-control group: OHI plus an EO mouthrinse (Listerine®)(3) test group: OHI plus the TCM mouthrinse (5% Fructus mume extract). Clinical examinations included Plaque Index (PI), Bleeding Index (BI) and Modified Gingival Index (MGI). Salivary microbial quantifications included total aerobic and anaerobic bacteria, Streptococci and Lactobacilli counts. Clinical and microbiological examinations were conducted at baseline, 3 and 6 months (T1, T2 and T3).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have at less 20 permanent teeth
* Subjects who have a healthy systemic condition
* Subjects with age range 13-35.
* Subjects who are no-smoker;
* Subjects who haven't taken antibiotic medicine within a 2 week period prior
* Subjects who do not currently undergo any medication or will undergo any medication in next six months
* Subjects who have not dental diseases that required ongoing treatment, which would confound the evaluation of result
* Subjects who are competent in giving consents
* Subjects who are not pregnant or lactating women
* Subjects who do not report teeth sensitivity
* Subjects who are not allergic to ethanol
* Subjects presented a minimum level of pre-existing gingivitis (MGI>1) but without peridontitis.(probing depth>4mm)

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Gingival index | 6 months
  Modified gingival index
Plaque index | 6 months
  plaque index
gingival bleeding index | 6 months
  gingival bleeding index

SECONDARY OUTCOMES:
Salivary cytokines | 6 months
  Salivary inflammatory cytokines (IL-1β and MIF) levels were detected by ELISA assay.
Adverse Events | 6 months
  the number of participants with side effects or adverse events were recorded throughout the whole study time.
Salivary bacteria counts | 6 months
  Salivary microbial quantifications included total aerobic and anaerobic bacteria, streptococci and lactobacilli counts.

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Wong, PhD, Principal Investigator — Faculty of Dentistry, The University of Hong Kong
Locations (1):
- Faculty of Dentistry, HKU, Hong Kong, China